CLINICAL TRIAL: NCT03479658
Title: Dose-effect of HIIT on Cardiovascular Health of Children Aged 9 to 10 Years Old Participating in a School Based Multidisciplinary Intervention Program: a Pilot Study
Brief Title: Dose-effect of HIIT on Cardiovascular Health of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pública de Navarra (Other)
Responsible Party: Principal Investigator, Idoia Labayen, Principal Investigator, Universidad Pública de Navarra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI-018/17
Record Dates: First submitted 2018-02-20; First posted 2018-03-27 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Cardiovascular Diseases Risk; Adiposity
Keywords: HIIT; nutritional education; Dose-effect; school; children; cardiovascular; adiposity; blood pressure; fitness
MeSH Terms: conditions — Obesity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIIT two sessions (Experimental): Two sessions per week of HIIT + nutritional education (1 session/week)
  Interventions: Behavioral: High intensity interval training; Behavioral: Nutritional education
- HIIT one session (Experimental): One session per week of HIIT + nutritional education (1 session/week)
  Interventions: Behavioral: High intensity interval training; Behavioral: Nutritional education
- Nutritional education (Active Comparator): Nutritional education (1 session/week)
  Interventions: Behavioral: Nutritional education

INTERVENTIONS:
Behavioral: High intensity interval training — Two schools with four classes/groups of 4th degree of children will participate in the pilot study (i.e., age of children 9-10 years old). One of them has two physical education (PE) sessions per week and the other has only one PE session per week. In the school with two PE sessions, two classes will be randomly assigned to HIIT (2 sessions/week) +nutrition group, and two to the nutrition group. Similarly, in the school with one PE session per week, two classes will be randomly assigned to HIIT (1 session/week) + nutrition and two classes to the nutrition goup. Both HIIT and nutritional education sessions will be integrated integrated into the physical education and sciences sessions of the schools. The duration of the intervention will be of eight weeks.
  Arms: HIIT one session; HIIT two sessions
Behavioral: Nutritional education — School-based nutritional education on healthy dietary habits

SUMMARY:
An adequate physical activity level has important effects on cardiovascular health of children. However, the scientific literature suggests that few children meet the physical activity recommendations to obtain these cardiovascular benefits which may have immediate and long term consequences in public health. High intensity interval training (HIIT) has emerged as an effective strategy for improving physical and mental health in children. To note that HIIT can be completed in a shorter period of time and its results in physical health seem to be equivalent to those obtained in longer sessions of traditional aerobic training. However, there is no information about the dose of HIIT needed to obtain significant effects on cardiovascular health of children.

The adoption of healthy dietary habits is also important in the prevention of obesity and cardiovascular diseases.

School-based programs including physical activity and nutritional education have been recommended as important components of programs aiming to prevent obesity and cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

All school children able to attend the physical education sessions of the school

-

Exclusion Criteria:

* Children with medical condition that limits physical activity

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Change in cardiorespiratory fitness | Change from baseline cardiorespiratory fitness at eight weeks
  20m shuttle run test (Alpha battery)

SECONDARY OUTCOMES:
Change in Body fat | Change from baseline body fat at eight weeks
  Body fat percent measured by bioimpedance
Change in Ankle-brachial index | Change from baseline Ankle-brachial index at eight weeks
  Automated simultaneous blood pressure measurement
Change in Dietary habits | Change from baseline Dietary habits at eight weeks
  Food frequency questionnaire and 24h recall
Change in Muscular strength | Change from baseline Muscular strength at eight weeks
  Handgrip strength and long jump (Alpha battery)
Change in speed-agility | Change from baseline speed agility at eight weeks
  4x10m speed agility test (Alpha battery)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Health Sciences, Universidad Pública de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No